CLINICAL TRIAL: NCT01049113
Title: Phase 1, Dose Escalation Study To Assess the Safety, Pharmacokinetics and Activity of 2-Hour Continuous Intravenous Dosing of ON 013105 Administered Weekly in Patients With Relapsed/Refractory Lymphoma and Acute Lymphoid Leukemia
Brief Title: Safety Study of ON 013105 in Lymphoma and Acute Lymphoid Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of available clinical drug supply
Sponsor: Traws Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ON-013105-01
Record Dates: First submitted 2010-01-11; First posted 2010-01-14 (Estimated); Last update posted 2015-12-08 (Estimated); Status verified 2015-12

CONDITIONS: Lymphoma; Acute Lymphocytic Leukemia
Keywords: Lymphoma; B-cell Acute Lymphocytic Leukemia; ALL
MeSH Terms: conditions — Lymphoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma | interventions — ON 013105

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ON 013105 (Experimental): ON 013105 administered intravenously as 2-hour infusion once a week for 3 weeks of 3-week cycles. This is dose escalation study; starting dose is 17 mg.
  Interventions: Drug: ON 013105

INTERVENTIONS:
Drug: ON 013105 — 2-hour intravenous infusion once a week. Starting dose is 17 mg. Maximum dose will be 1525 mg.
  Other Names: briciclib

SUMMARY:
This is an open-label, dose-escalation Phase 1 study of the investigational agent, ON 013105. In laboratory animal studies, ON 013105 has demonstrated anti-cancer activity. The purpose of this study is to determine the highest dose of ON 013105 that can be given safely in patients with relapsed/refractory Lymphoma or B-cell Acute Lymphocytic Leukemia (Philadelphia chromosome negative). Patients will receive weekly 2-hour IV infusions of ON 013105 at higher and higher doses until intolerable side effects are observed. It is important to know the highest safe dose so additional studies can be done.

DETAILED DESCRIPTION:
This is an open-label, dose-escalation Phase I study of ON 013105 in patients with relapsed/refractory Lymphoma or B-cell Acute Lymphocytic Leukemia (Philadelphia chromosome negative) who have satisfied all inclusion/exclusion criteria. Patients will receive weekly 2-hour IV infusions of ON 013105, until evidence of disease progression, intolerable adverse events, or withdrawal of patient consent. Up to 12 additional patients will be treated at the RPTD level. The starting dose will be 17 mg over a 2-hour weekly infusion. Each cycle will comprise three weeks.

Up to 43 patients may be enrolled, of which approximately 7 to 37 patients will be enrolled in the dose escalation portion of the study to determine the RPTD. After the maximally administered dose is attained and at least six patients have received a tentative RPTD, up to 6 additional patients may be enrolled in the dose confirmation phase to confirm the RPTD level.

Treatment will be administered in the Clinical Research center for the first dose for all patients at each given dose level. If there is no toxicity, then subsequent doses at that level for that patient may be administered on an outpatient basis, unless hospitalization is required for another reason.

According to the Simon accelerated titration design, one-patient cohorts and 100% dose increments will be implemented until non-hematological grade 2 toxicity is observed during the first 3-week cycle. The design will then convert to standard 3/6 patient cohorts starting at the dose level where grade 2 toxicity was observed and following 40% dose increments for the subsequent cohorts.

If none of the first three patients experiences a dose-limiting toxicity (DLT) during the first cycle (3 weeks), the next 3 patients will receive the next dose level. If there is a DLT in one of the first three patients, this dose level will be expanded to 6 patients. If 1 patient out of 6 experiences DLT, the next patients will receive the next dose level. If ≥ 2 patients experience DLT at any dose level, this dose level will be declared the Maximally Administered Dose. The Maximally Tolerated Dose (MTD) and RPTD will be the highest dose level below the Maximally Administered Dose with 0 out of 3 patients or one out of 6 patients with DLT. Dosing will be reduced to the immediate lower dose for any patient who experiences a DLT at any time.

If Grade 1 non-hematological toxicity occurs, treatment will be continued at the original dose without dose reduction.

Patients with stable disease or response can continue treatment up to eight 3-week cycles. Further continuation will be determined by the clinical judgment of the Investigator. Patients who drop out for any reason may not re-enter the trial.

Blood samples will be collected during Day 1 of the first cycle for pharmacokinetic assessment. Responses will be assessed according to Cheson, B.D., et al., Revised Response Criteria for Malignant Lymphoma, J Clin Oncol 2007. 25: p. 579-86.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Documented (cytologically confirmed) relapsed/ refractory Lymphoma or B-cell Acute Lymphocytic Leukemia (Philadelphia chromosome negative)
* ECOG Performance Status score of 0, 1, or 2 (see Attachment 1)
* Expected survival, in the opinion of the Investigator, of at least 3 months, to allow a sufficient observation period for evaluation of ON 013105
* Recovery to at least grade I from adverse effects of prior therapies
* Adequate contraceptive [including prescription oral contraceptives (birth control pills), contraceptive injections, intrauterine device (IUD), double-barrier method (spermicidal jelly or foam with condoms or diaphragm), contraceptive patch, or surgical sterilization] before entry and throughout the study for female patients of reproductive potential
* Female patient with reproductive potential must have a negative serum beta-HCG pregnancy test at screening
* Willing to adhere to the prohibitions and restrictions specified in this protocol
* Patient (or his/her legally authorized representative) must have signed an informed consent document indicating that he/she understands the purpose of and procedures required for the study and is willing to participate in the study

Exclusion Criteria:

* Grade 3 thrombocytopenia (platelets <50,000/µL) or neutropenia (ANC <1000/µL) ) except if documented evidence of bone marrow involvement of lymphoma or leukemia contributing to cytopenias.
* Any active malignancy within the past year except basal cell or squamous cell skin cancer or carcinoma in situ of the cervix or breast
* History of HIV-1 seropositivity
* Uncontrolled intercurrent illness including, but not limited to symptomatic congestive heart failure, unstable angina pectoris or cardiac arrhythmia
* Active infection not adequately responding to appropriate therapy.
* Total bilirubin > 1.5 mg/dL not related to hemolysis or Gilbert's disease, AST/ALT > 1.5 X ULN
* Serum creatinine > 1.5 mg/dL or calculated creatinine clearance < 60 ml/min.
* Ascites requiring active medical management including paracentesis, or hyponatremia (defined as serum sodium value of <130 Meq/L).
* Women patients who are pregnant or lactating
* Male patients with female sexual partners who are unwilling to follow the strict contraception requirements described in this protocol (see Section 4.4).
* Major surgery without full recovery or major surgery within 3 weeks of ON 013105 treatment start.
* Uncontrolled hypertension (defined as a systolic pressure ³ 180 and/or a diastolic pressure ³ 110)
* New onset seizures (within 3 months prior to the first dose of ON 013105) or poorly controlled seizures
* Any concurrent investigational agent or chemotherapy, radiotherapy or immunotherapy
* Psychiatric illness/social situations that would limit the patient's ability to tolerate and/or comply with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2009-11; Primary Completion 2014-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Safety based on adverse events, hematology and chemical laboratory values, urinalysis, coagulation, ECG, vital signs, physical examination. | 2 years

SECONDARY OUTCOMES:
Tumor response (according to Cheson, B.D., et al., Revised Response Criteria for Malignant Lymphoma, J Clin Oncol 2007. 25: p. 579-86). | 2 years
Non-compartmental pharmacokinetic analysis of drug concentrations in plasma including area under concentration time curve, half-life, clearance. | Day 1 of first cycle

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Cultrera, MD, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida, United States

REFERENCES:
- [Background] Park IW, Reddy MV, Reddy EP, Groopman JE. Evaluation of novel cell cycle inhibitors in mantle cell lymphoma. Oncogene. 2007 Aug 16;26(38):5635-42. doi: 10.1038/sj.onc.1210350. Epub 2007 Mar 19. PMID 17369860
- [Background] Prasad A, Park IW, Allen H, Zhang X, Reddy MV, Boominathan R, Reddy EP, Groopman JE. Styryl sulfonyl compounds inhibit translation of cyclin D1 in mantle cell lymphoma cells. Oncogene. 2009 Mar 26;28(12):1518-28. doi: 10.1038/onc.2008.502. Epub 2009 Feb 9. PMID 19198627
- See also: The Leukemia & Lymphoma Society — http://www.leukemia-lymphoma.org